CLINICAL TRIAL: NCT06666296
Title: Sustainable Eating for a Healthy Tomorrow - Effectiveness of Digital Nutrition Workshops to Implement the Planetary Health Diet for Hospital Employees
Acronym: EatGood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Deutsche Bundesstiftung Umwelt (Unknown)
Responsible Party: Principal Investigator, Heidemarie Haller, Director of Research, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 24-11823-BO
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Personnel, Hospital; Healthy Volunteers
MeSH Terms: interventions — Media Exposure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The following digital measures are used to provide employees in the intervention group with comprehensive information at various levels and to create a sense of belonging: A digital recipe collection, an email newsletter, digital/hybrid teaching kitchen events and digital cafés with expert input and discussion groups. In addition, participants are provided with interesting information via the hospital's Instagram account and are constantly reminded of the campaign. When selecting the digital media, emphasis was placed on integrating different learning methods. Through self-learning content, such as the email newsletter, participants can absorb the information at their own pace, make a connection and evaluate it. The topics are then explored and discussed in greater depth in digital events. Individual priorities can be set in group discussions. Through regular input, participants experience a growth phase.
  Interventions: Behavioral: Digital collection of recipes; Behavioral: E-Mail-Newsletter; Behavioral: digital/hybrid teaching kitchen; Behavioral: Digital events (digital cafés); Behavioral: Social-Media
- Control group (Other): The control group will have access to the digital prescription collection, which is being developed on the basis of the Planetary Health Diet. In addition, the control group can use information on the clinic's Instagram account. In addition to access to the above-mentioned recipes and information via the Instagram channel, the intervention group receives additional digital support.
  Interventions: Behavioral: Digital collection of recipes; Behavioral: Social-Media

INTERVENTIONS:
Behavioral: Digital collection of recipes — The digital recipe collection is created for private use. This collection contains recipes for every meal of the day to ensure a Planetary Health Diet throughout the day. This includes digital weekly plans with corresponding dishes, including shopping lists, to simplify implementation in everyday life. This enables participants to make quick meal choices and simplify their shopping. Employees are encouraged to use this digital recipe collection to prepare their meals over a defined period of time. In addition, the kitchen management of the university hospital will be asked to assist with the creation of the recipes. The project benefits from the experience of the kitchen staff. Popular recipes can be used across projects.
Behavioral: E-Mail-Newsletter — The e-mail newsletter contains information on the Planetary Health Diet (background, urgency, goals, etc.). Regular contact by e-mail enables a fast, uncomplicated and personal exchange with the participants, uncomplicated and personal exchange with the participants. The e-mail support encourages participants to actively engage with the topic. The newsletter is supplemented by instructional kitchen videos (one person cooks a recipe from the recipe collection), checklists (e.g. "How sustainable am I already acting?"), tasks (e.g. three possible measures for a more sustainable diet) or food information (e.g. seasonal plan for fruit and vegetables). This provides participants with important information at regular intervals and ensures compliance.
  Arms: Intervention group
Behavioral: digital/hybrid teaching kitchen — Recipes, cooking techniques, shopping tips and recommendations for implementing the Planetary Health Diet are taught in the digital/hybrid teaching kitchen. The focus here is on fun, good taste and interesting experiences. A shared experience can be created through such cooking events. The teaching kitchen events can be supplemented by the participation of the kitchen management in order to benefit from their special cooking skills and wealth of experience. The positive aspect of the digital training kitchen is the easy access to information, as this does not have to be read, but is conveyed visually.
  Arms: Intervention group
Behavioral: Digital events (digital cafés) — Events are planned that will be set up via the "digital café" for in-depth discussions and exchanges about the content. Fixed dates are planned at which the study participants can meet digitally. In this protected setting, the topics of the study will be discussed in a convivial atmosphere. The personal exchange enables a deeper examination of the topic. The online events give participants the opportunity to interact directly with the study coordinators and other participants in order to effectively and sustainably change the participants' perception and awareness of sustainable nutrition through the various intervention points.
  Arms: Intervention group
Behavioral: Social-Media — A dedicated Instagram account for this project will be created for the center, where valuable content on the Planetary Health Diet will be shared regularly. The test subjects can also use this platform to exchange information.

SUMMARY:
The investigators will explore the effect of digital media on communicating a planetary diet and invite participants to change dietary habits. Standardized questionnaires, physical examinations, and qualitative interviews will be used to obtain data on the effectiveness of the intervention. Once initial assessments are complete, a blinded researcher will randomly assign participants to one of two groups, without influence from either participants or study coordinators.

Both groups will participate in a nutrition course over a 13-week period, followed by a booster session five months after randomization, and will be encouraged to practice the methods at home. One group will receive intensive support, including a digital training program (around 2 hours per week), while the other group will receive digital information and sustainable recipes with limited support (about 30 minutes per week).

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 years
* Employee at the University Hospital Essen
* A functioning smartphone
* Moderate willingness (at least 5 points on NRS) to want to change diet
* Access to digital media and social media

Exclusion Criteria:

* Insufficient knowledge of the German language
* Simultaneous participation in other clinical intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2025-08-12 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
Healthy Eating Habits - Healthy Plant-based Diet Index (hPDI) | Month 3
  Changes in heathy eating habits are measured using a generally recognized Food Frequency Questionnaire (FFQ) in the validated German DEGS-Version from the Robert Koch Institute, Germany. The DEGS comprises 53 questions and records the frequency of consumption of various food groups and drinks over a certain period of time. The following habits are assessed: healthy plant-based foods, less healthy plant-based foods and animal-based foods. The Helathy Plant-based Diet Index (hPDI) is calculated from the DEGS questionnaire. The score of the hPDI can range from 18 to 90, with a higher index reflecting a more plant-based and less animal-based diet.

SECONDARY OUTCOMES:
Healthy Eating Habits - Healthy Plant-based Diet Index (hPDI) | Month 6
  Changes in heathy eating habits are measured using a generally recognized Food Frequency Questionnaire (FFQ) in the validated German DEGS-Version from the Robert Koch Institute, Germany. The DEGS comprises 53 questions and records the frequency of consumption of various food groups and drinks over a certain period of time. The following habits are assessed: healthy plant-based foods, less healthy plant-based foods and animal-based foods. The Helathy Plant-based Diet Index (hPDI) is calculated from the DEGS questionnaire. The score of the hPDI can range from 18 to 90, with a higher index reflecting a more plant-based and less animal-based diet.
Willingness to Change (PIAC) | Month 3
  The questionnaire PIAC (Perception, intention and ability for change) questionnaire relates to the ability to change health behavior, habits and living conditions. The statements are based on respondents' experiences and cover various factors such as substance use, dietary habits, lack of exercise and disease-promoting behaviors. The PIAC contains 13 questions that can be answered at a scale from "strongly disagree" (0 points) to "strongly agree" (4 points). A higher score (0-52 range) shows a positive attitude, strong intent, and ability to adopt healthier behaviors.
Willingness to Change (PIAC) | Month 6
  The questionnaire PIAC (Perception, intention and ability for change) questionnaire relates to the ability to change health behavior, habits and living conditions. The statements are based on respondents' experiences and cover various factors such as substance use, dietary habits, lack of exercise and disease-promoting behaviors. The PIAC contains 13 questions that can be answered at a scale from "strongly disagree" (0 points) to "strongly agree" (4 points). A higher score (0-52 range) shows a positive attitude, strong intent, and ability to adopt healthier behaviors.
Adaptive Coping with Disease (AKU) | Month 3
  The questionnaire AKU (AKU is an acronym of the German translation of "Adaptive Coping with Disease") meassures active and adaptive behaviors to maintain health. It offers the opportunity to record and quantify the implementation of strategies to promote health in different contexts, taking into account both external influences and individual, internal convictions. We used one subsclae of the AKU (Conscious way of living), which consists of 5 questions and ranges from "Does not apply at all" (0 points) to "Applies exactly" (4 points). Therefore, the sum score ranges from 0-20. A high score indicates strong adaptive health behavior and good implementation of health-promoting strategies.
Adaptive Coping with Disease (AKU) | Month 6
  The questionnaire AKU (AKU is an acronym of the German translation of "Adaptive Coping with Disease") meassures active and adaptive behaviors to maintain health. It offers the opportunity to record and quantify the implementation of strategies to promote health in different contexts, taking into account both external influences and individual, internal convictions. We used one subsclae of the AKU (Conscious way of living), which consists of 5 questions and ranges from "Does not apply at all" (0 points) to "Applies exactly" (4 points). Therefore, the sum score ranges from 0-20. A high score indicates strong adaptive health behavior and good implementation of health-promoting strategies.
Self-efficacy (HSSES) | Month 3
  Health-specific self-efficacy scale (HSSES) meassures the confidence in the ability to accomplish certain health tasks, even if they are challenging. In the area of nutrition, self-efficacy can positively influence an intervention. HSSES is a set of 5 questions to be answered on a scale of 0-4: (0) very uncertain, (1) somewhat uncertain, (2) I cannot say, (3) somewhat certain, and (4) very certain. Therefore, the sum ranges between 0-20. A higher score on the HSSES indicates strong confidence in one's ability to change their diet, which can positively influence behavior.
Self-efficacy (HSSES) | Month 6
  Health-specific self-efficacy scale (HSSES) meassures the confidence in the ability to accomplish certain health tasks, even if they are challenging. In the area of nutrition, self-efficacy can positively influence an intervention. HSSES is a set of 5 questions to be answered on a scale of 0-4: (0) very uncertain, (1) somewhat uncertain, (2) I cannot say, (3) somewhat certain, and (4) very certain. Therefore, the sum ranges between 0-20. A higher score on the HSSES indicates strong confidence in one's ability to change their diet, which can positively influence behavior.
Quality of Life (WHO-5) | Month 3
  The WHO-5 Index (Well-being index of the WHO) is a self-assessment method for measuring quality of life. Participants answers 5 questions on a six-point Likert scale (from 0 = "At no time" to 5 = "All the time"). The sum score is calculated by adding up the 5 item values, with higher values indicating better quality of life. Therefore, a score to be achieved is between 0-25.
Quality of Life (WHO-5) | Month 6
  The WHO-5 Index (Well-being index of the WHO) is a self-assessment method for measuring quality of life. Participants answers 5 questions on a six-point Likert scale (from 0 = "At no time" to 5 = "All the time"). The sum score is calculated by adding up the 5 item values, with higher values indicating better quality of life. Therefore, a score to be achieved is between 0-25.
Environmental and Climate Behavior (YCSCB) | Month 3
  The YCSCB (Young Consumers' Sustainable Consumption Behavior) scale is used to meassure the respondent's sustainable consumption behavior. The questionnaire contains 14 short questions that can be answered in four categories: "never" (0 points), "sometimes" (1 points), "often" (2 points) and "always" (3 points). Therefore, a score between 0-51 points can be achieved. A higher score on the YCSCB indicates a strong sustainable behavior.
Environmental and Climate Behavior (YCSCB) | Month 6
  The YCSCB (Young Consumers' Sustainable Consumption Behavior) scale is used to meassure the respondent's sustainable consumption behavior. The questionnaire contains 14 short questions that can be answered in four categories: "never" (0 points), "sometimes" (1 points), "often" (2 points) and "always" (3 points). Therefore, a score between 0-51 points can be achieved. A higher score on the YCSCB indicates a strong sustainable behavior.
Body Mass Index (BMI) | Month 3
  The measurement of body weight is a fundamental indicator of overall health and can provide insights into potential health risks. Increased body weight and therefore Body Mass Index (BMI) may indicate overweight or obesity, which is associated with a higher risk of various diseases, including cardiovascular diseases, diabetes, and metabolic syndrome. Regular weight monitoring allows for the early detection of changes in body weight, enabling the implementation of preventive measures if necessary. Body weight is therefore measured on a calibrated and validated scale, while wearing only underwear. BMI ranges are categorized as follows: underweight: <18.5, normal weight: 18.5-24.9, overweight: 25-29.9, obesity: ≥30.
Body Mass Index (BMI) | Month 6
  The measurement of body weight is a fundamental indicator of overall health and can provide insights into potential health risks. Increased body weight and therefore Body Mass Index (BMI) may indicate overweight or obesity, which is associated with a higher risk of various diseases, including cardiovascular diseases, diabetes, and metabolic syndrome. Regular weight monitoring allows for the early detection of changes in body weight, enabling the implementation of preventive measures if necessary. Body weight is therefore measured on a calibrated and validated scale, while wearing only underwear. BMI ranges are categorized as follows: underweight: <18.5, normal weight: 18.5-24.9, overweight: 25-29.9, obesity: ≥30.
Body weight | Month 3
  Body weight measurement is a fundamental indicator of overall health and can provide valuable insights into potential health risks. A persistent increase in body weight can indicate overweight or obesity, which are associated with an elevated risk of various diseases, including cardiovascular diseases, diabetes, and metabolic disorders. Conversely, unintended weight loss may point to underlying health issues such as malnutrition or chronic illness. Regular monitoring of body weight allows for early detection of such changes, supporting timely preventive or therapeutic interventions. Body weight is measured using a calibrated and validated scale, while the participant wears only underwear.
Body weight | Month 6
  Body weight measurement is a fundamental indicator of overall health and can provide valuable insights into potential health risks. A persistent increase in body weight can indicate overweight or obesity, which are associated with an elevated risk of various diseases, including cardiovascular diseases, diabetes, and metabolic disorders. Conversely, unintended weight loss may point to underlying health issues such as malnutrition or chronic illness. Regular monitoring of body weight allows for early detection of such changes, supporting timely preventive or therapeutic interventions. Body weight is measured using a calibrated and validated scale, while the participant wears only underwear
Waist Circumference | Month 3
  The measurement of waist circumference plays a crucial role in assessing the risk of metabolic syndrome and current health status. By determining waist circumference, the distribution of body fat and the mass of visceral fat (abdominal fat) can be evaluated, enabling an individual risk assessment of concomitant diseases. Abdominal obesity, characterized by an increased proportion of visceral fat, is associated with a higher risk of metabolic and cardiovascular health issues. Waist measurement is independent of body size and offers insights into intra-abdominal fat mass and total body fat. Women: low risk: <80 cm, increased risk: 80-88 cm, highly increased risk: >88 cm. Men: low risk: <94 cm, increased risk: 94-102 cm, highly increased risk.
Waist Circumference | Month 6
  The measurement of waist circumference plays a crucial role in assessing the risk of metabolic syndrome and current health status. By determining waist circumference, the distribution of body fat and the mass of visceral fat (abdominal fat) can be evaluated, enabling an individual risk assessment of concomitant diseases. Abdominal obesity, characterized by an increased proportion of visceral fat, is associated with a higher risk of metabolic and cardiovascular health issues. Waist measurement is independent of body size and offers insights into intra-abdominal fat mass and total body fat. Women: low risk: <80 cm, increased risk: 80-88 cm, highly increased risk: >88 cm. Men: low risk: <94 cm, increased risk: 94-102 cm, highly increased risk.
Adverse events (AEs) | Month 0 to 3 (during intervention)
  Safety was operationalized as the number of (participants with) adverse events (AE) or study withdrawals due to AEs. AEs were defined as any untoward medical occurrence in a participant, which did not have to have a defined causal relationship with the treatment being studied. Cases of any untoward medical occurrence that, at any dose, resulted in death, were life-threatening, required inpatient hospitalization, or caused persistent or significant disability were assessed as serious AEs.

OTHER OUTCOMES:
Work Engagement (UWES) | Month 0
  Work engagement is collected through the questionnaire UWES (Utrecht Work Engagement Scale). Work engagement is considered to be the supposed opposite of burnout. This is because, unlike people who suffer from burnout, engaged employees have a sense of energized and effective connection to their work activities and see themselves as being able to cope well with the demands of their job. The questionnaire contains nine questions to be answered on a scale of 0-6. This means that you can achieve a score between 0-54. A high score (40-54) on the UWES indicates strong work energy, commitment and effectiveness, which indicates a low risk of burnout. Low scores (0-18) indicate low engagement and potential burnout.
Work Engagement (UWES) | Month 3
  Work engagement is collected through the UWES (Utrecht Work Engagement Scale). Work engagement is considered to be the supposed opposite of burnout. This is because, unlike people who suffer from burnout, engaged employees have a sense of energized and effective connection to their work activities and see themselves as being able to cope well with the demands of their job. The questionnaire contains nine questions to be answered on a scale of 0-6. Therefore, a score between 0-54 can be achieved. A high score on the UWES indicates strong work energy, commitment and effectiveness, which indicates a low risk of burnout.
Work Engagement (UWES) | Month 6
  Work engagement is collected through the UWES (Utrecht Work Engagement Scale). Work engagement is considered to be the supposed opposite of burnout. This is because, unlike people who suffer from burnout, engaged employees have a sense of energized and effective connection to their work activities and see themselves as being able to cope well with the demands of their job. The questionnaire contains nine questions to be answered on a scale of 0-6. Therefore, a score between 0-54 can be achieved. A high score on the UWES indicates strong work energy, commitment and effectiveness, which indicates a low risk of burnout.
Workload (NRS) | Month 0
  Workload is measured using an NRS (Numeric Rating Scale). A high workload can reduce adherence to the intervention and lead to stress or burnout. Therefore, it is important to ensure that the intervention can be realistically integrated into participants' daily lives and that appropriate support is provided. Therefore, the following question is asked: Please use the scale to indicate how much stress you currently feel as a result of your work. The scale ranges from 0% (0 points) to 100% (10 points) in eleven steps. A high score on the NRS indicates a heavy workload and increased risk of stress.
Workload (NRS) | Month 3
  Workload is measured using an NRS (Numeric Rating Scale). A high workload can reduce adherence to the intervention and lead to stress or burnout. Therefore, it is important to ensure that the intervention can be realistically integrated into participants' daily lives and that appropriate support is provided. Therefore, the following question is asked: Please use the scale to indicate how much stress you currently feel as a result of your work. The scale ranges from 0% (0 points) to 100% (10 points) in eleven steps. A high score on the NRS indicates a heavy workload and increased risk of stress.
Workload (NRS) | Month 6
  Workload is measured using an NRS (Numeric Rating Scale). A high workload can reduce adherence to the intervention and lead to stress or burnout. Therefore, it is important to ensure that the intervention can be realistically integrated into participants' daily lives and that appropriate support is provided. Therefore, the following question is asked: Please use the scale to indicate how much stress you currently feel as a result of your work. The scale ranges from 0% (0 points) to 100% (10 points) in eleven steps. A high score on the NRS indicates a heavy workload and increased risk of stress.
Mental Well-Being (PHQ-4) | Month 0
  The PHQ-4 questionnaire (Patient Health Questionaire) is used to assess mental well-being.The questionnaire consists of four questions and a four-point scale from 0 till 3. The PHQ-4 can achieve a score between 0-12. A higher score on the PHQ-4 indicates significant mental stress, which could make it difficult to implement an intervention.
Mental Well-Being (PHQ- 4) | Month 3
  The PHQ-4 questionnaire (Patient Health Questionaire) is used to assess mental well-being.The questionnaire consists of four questions and a four-point scale from 0 till 3. The PHQ-4 can achieve a score between 0-12. A higher score on the PHQ-4 indicates significant mental stress, which could make it difficult to implement an intervention.
Mental Well-Being (PHQ- 4) | Month 6
  The PHQ-4 questionnaire (Patient Health Questionaire) is used to assess mental well-being.The questionnaire consists of four questions and a four-point scale from 0 till 3. The PHQ-4 can achieve a score between 0-12. A higher score on the PHQ-4 indicates significant mental stress, which could make it difficult to implement an intervention.
Client Satisfaction Questionnaire (CSQ) | Month 3
  Satisfaction with the intervention is meassured directly after completion of the intervention. The CSQ (Client Satisfaction Questionnaire) uses eight items to measure general satisfaction with various aspects of the treatment received. The items are scored from 1 (most unfavorable) to 4 (most positive) according to their polarity and added up to an overall score ranged 8-32 with higher scores indicate higher satisfaction. .
Expectation of Treatment Effectiveness (NRS) | Month 0
  The expectation of treatment effectiveness is meassured by an NRS using two questions. The first question: "At this point in time, how successful do you think this course will be in improving the quality of your functioning?" ranges from not at all (0) to very useful (10) and the second question: "At the end of the course, how much improvement in your functioning do you think you will actually experience?" ranges from 0% (0) to 100% (10). A higher score indicates optimistic expectations of treatment success.
Compliance (Diary) | Month 0 to 3 (during intervention)
  Two questions are integrated into the study diary to record the daily dietary behavior of the test subjects using a Likert scale: "Please indicate to what extent you managed to eat the 5 recommended servings of fruits and vegetables today" and: "Please indicate to what extent you managed to eat servings of fruits and vegetables today, specifically the 1 recommended serving of legumes."

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Integrative Medicine and Planetary Health, University Hospital Essen, University of Duisburg-Essen, Essen, Germany

IPD SHARING:
Plan to Share IPD: No